CLINICAL TRIAL: NCT00696280
Title: Observational Study of Delayed Nausea and Vomiting Following Administration of Carboplatin Containing Regimens for Treatment of Cancer
Brief Title: Observational Study of Delayed Nausea and Vomiting
Acronym: DelayedNaus
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 06-0981 / 201104043
Record Dates: First submitted 2008-06-09; First posted 2008-06-12 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-06

CONDITIONS: Vomiting
Keywords: nausea; vomiting; Carboplatin; cancer; delayed emesis following treatment with carboplatin
MeSH Terms: conditions — Vomiting; Nausea; Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: All patients will be given the Functional Living Index - Emesis (FLIE) standardized questionnaire during their scheduled clinic visit prior to receiving chemotherapy.
  This is a self-administered questionnaire. Patients will complete the questionnaire during the 5 days following carboplatin administration (at 24 hours, 48 hours, 72 hours, and 96 hours) of their first and third cycles of chemotherapy.
  Patients will also be interviewed by a trained CRA or research nurse over the telephone 24-48 hours following carboplatin administration in order to assess the severity of the delayed nausea and vomiting.
  Interventions: Behavioral: Functional Living Index - Emesis

INTERVENTIONS:
Behavioral: Functional Living Index - Emesis

SUMMARY:
Delayed emesis following administration of carboplatin-based chemotherapy despite prophylaxis with standard antiemetic prophylaxis (5-HT3 and corticosteroid) remains a clinically significant and distressing problem for patients with cancer. The incidence of delayed emesis appears to be higher in women compared to men.

DETAILED DESCRIPTION:
All patients will be given the Functional Living Index- Emesis (FLIE), a standardized questionnaire. This is a self-administered questionnaire to assess the impact of nausea and vomiting on the patient's functional living, including physical activities, social and emotional function, and ability to enjoy food and drink. Patients will complete the questionnaire during the 5 days following carboplatin administration (at 24 hours, 48 hours, 72 hours and 96 hours) during their first and third cycles of chemotherapy. The questionnaire should take approximately 10 minutes or less to complete.

Patients will also be interviewed by a trained CRA or research nurse over the telephone 24-48 hours following carboplatin administration in order to assess the severity of the delayed nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have newly diagnosed, histologically or cytologically proven cancer, and be scheduled to receive chemotherapy with carboplatin at AUC 5 or above.
* Patients should receive standard antiemetic prophylaxis prior to carboplatin administration, defined as 5-HT3 antagonist and dexamethasone. We will include only patients whose standard care includes treatment with a carboplatin-containing regimen and who are not being treated with aprepitant (Emend®).
* Age >= 18.
* After being informed of the treatment involved, patients must give written consent.
* Entry to this study is open to both men and women and to all racial and ethnic subgroups.

Exclusion Criteria:

* No prior cytotoxic chemotherapy within the last 5 years.
* Should not be pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have received one treatment of carboplatin
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2006-11; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Characterize the incidence of delayed emesis following administration of carboplatin-containing chemotherapy regimens | After 1st cycle of chemotherapy
  Despite appropriate administration of standard 5-HT3 receptor antagonist antiemetic prophylaxis after the first cycle of chemotherapy.

SECONDARY OUTCOMES:
Characterize the incidence of delayed emesis following administration of carboplatin-containing chemotherapy regimens | After 3rd cycle of chemotherapy
  Despite appropriate administration of standard antiemetic prophylaxis after the third cycle of chemotherapy
Characterize the differences in incidence of delayed nausea and vomiting among male and female patients receiving carboplatin. | Through the end of 3 cycles of therapy
Assess the need for breakthrough nausea and vomiting control in patients following administration of carboplatin-containing chemotherapy regimens | Through the end of 3 cycles of therapy
  Despite appropriate administration of standard antiemetic prophylaxis.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Q Baggstrom, M.D., Principal Investigator — Washington University School of Mecicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Kris MG, Gralla RJ, Clark RA, Tyson LB, O'Connell JP, Wertheim MS, Kelsen DP. Incidence, course, and severity of delayed nausea and vomiting following the administration of high-dose cisplatin. J Clin Oncol. 1985 Oct;3(10):1379-84. doi: 10.1200/JCO.1985.3.10.1379. PMID 4045527
- [Background] Ettinger D, Johnson B. Update: NCCN small cell and non-small cell lung cancer Clinical Practice Guidelines. J Natl Compr Canc Netw. 2005 Nov;3 Suppl 1:S17-21. No abstract available. PMID 16280105
- [Background] Raby B, Pater J, Mackillop WJ. Does knowledge guide practice? Another look at the management of non-small-cell lung cancer. J Clin Oncol. 1995 Aug;13(8):1904-11. doi: 10.1200/JCO.1995.13.8.1904. PMID 7636532
- [Background] Hesketh PJ, Kris MG, Grunberg SM, Beck T, Hainsworth JD, Harker G, Aapro MS, Gandara D, Lindley CM. Proposal for classifying the acute emetogenicity of cancer chemotherapy. J Clin Oncol. 1997 Jan;15(1):103-9. doi: 10.1200/JCO.1997.15.1.103. PMID 8996130
- [Background] du Bois A, Vach W, Kiechle M, Cramer-Giraud U, Meerpohl HG. Pathophysiology, severity, pattern, and risk factors for carboplatin-induced emesis. Oncology. 1996 Jun;53 Suppl 1:46-50. doi: 10.1159/000227640. PMID 8692551
- [Background] Delayed emesis induced by moderately emetogenic chemotherapy: do we need to treat all patients? The Italian Group for Antiemetic Research. Ann Oncol. 1997 Jun;8(6):561-7. PMID 9261525
- [Background] Hesketh PJ, Grunberg SM, Gralla RJ, Warr DG, Roila F, de Wit R, Chawla SP, Carides AD, Ianus J, Elmer ME, Evans JK, Beck K, Reines S, Horgan KJ; Aprepitant Protocol 052 Study Group. The oral neurokinin-1 antagonist aprepitant for the prevention of chemotherapy-induced nausea and vomiting: a multinational, randomized, double-blind, placebo-controlled trial in patients receiving high-dose cisplatin--the Aprepitant Protocol 052 Study Group. J Clin Oncol. 2003 Nov 15;21(22):4112-9. doi: 10.1200/JCO.2003.01.095. Epub 2003 Oct 14. PMID 14559886
- [Background] Poli-Bigelli S, Rodrigues-Pereira J, Carides AD, Julie Ma G, Eldridge K, Hipple A, Evans JK, Horgan KJ, Lawson F; Aprepitant Protocol 054 Study Group. Addition of the neurokinin 1 receptor antagonist aprepitant to standard antiemetic therapy improves control of chemotherapy-induced nausea and vomiting. Results from a randomized, double-blind, placebo-controlled trial in Latin America. Cancer. 2003 Jun 15;97(12):3090-8. doi: 10.1002/cncr.11433. PMID 12784346
- [Background] Lindley CM, Hirsch JD, O'Neill CV, Transau MC, Gilbert CS, Osterhaus JT. Quality of life consequences of chemotherapy-induced emesis. Qual Life Res. 1992 Oct;1(5):331-40. doi: 10.1007/BF00434947. PMID 1299465
- [Background] Martin AR, Pearson JD, Cai B, Elmer M, Horgan K, Lindley C. Assessing the impact of chemotherapy-induced nausea and vomiting on patients' daily lives: a modified version of the Functional Living Index-Emesis (FLIE) with 5-day recall. Support Care Cancer. 2003 Aug;11(8):522-7. doi: 10.1007/s00520-003-0482-4. Epub 2003 Jun 25. PMID 12827483
- [Background] Schipper H, Clinch J, McMurray A, Levitt M. Measuring the quality of life of cancer patients: the Functional Living Index-Cancer: development and validation. J Clin Oncol. 1984 May;2(5):472-83. doi: 10.1200/JCO.1984.2.5.472. PMID 6374052
- [Background] Martin AR, Carides AD, Pearson JD, Horgan K, Elmer M, Schmidt C, Cai B, Chawla SP, Grunberg SM. Functional relevance of antiemetic control. Experience using the FLIE questionnaire in a randomised study of the NK-1 antagonist aprepitant. Eur J Cancer. 2003 Jul;39(10):1395-401. doi: 10.1016/s0959-8049(03)00299-5. PMID 12826042
- [Result] Schnell FM. Chemotherapy-induced nausea and vomiting: the importance of acute antiemetic control. Oncologist. 2003;8(2):187-98. doi: 10.1634/theoncologist.8-2-187. PMID 12697943
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu